CLINICAL TRIAL: NCT06217666
Title: A Phase 1, Prospective, Standard Dose Escalation Study Examining the Safety and Toxicity of Stereotactic Body Radiotherapy (SBRT) Followed by PCX12 Immunotherapy Delivered by Intratumoral Injection for the Treatment of Patients With Locally Advanced Pancreatic Adenocarcinoma (LAPC)
Brief Title: Study Examining the Safety and Toxicity of Stereotactic Body Radiotherapy (SBRT) Followed by PCX12 Immunotherapy Delivered by Intratumoral Injection for the Treatment of Patients With Locally Advanced Pancreatic Adenocarcinoma (LAPC)
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Haoming (Carl) Qiu (Other)
Responsible Party: Sponsor-Investigator, Haoming (Carl) Qiu, Associate Professor - Department of Radiation Oncology (SMD), University of Rochester
Organization: University of Rochester (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: URGIP24061
Record Dates: First submitted 2024-01-09; First posted 2024-01-22 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Pancreatic Adenocarcinoma
Keywords: Pancreatic Adenocarcinoma; Pancreatic Cancer; PCX12; IL-12
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- PCX-12 (Experimental): PCX-12 is an experimental immunotherapy drug that is injected into the pancreatic cancer one time in attempt to stimulate the patient's immune system to fight the cancer.
  Interventions: Drug: PCX-12

INTERVENTIONS:
Drug: PCX-12 — treatment combining radiation therapy with PCX12

SUMMARY:
The purpose of this study is to determine whether a new treatment combining radiation therapy with PCX12 is safe and tolerable.

DETAILED DESCRIPTION:
Single center, open label, escalating dosage of PCX12 with standard of care practice for subjects who are diagnosed with adenocarcinoma of the head of the pancreas. Subjects with undergo standard of care radiation therapy and then start on PCX12 therapy starting at 200 ng/kg of PCX12 escalating to a potential maximum dosage of 800 ng/kg of PCX12 with adjacent tolerability and safety guidelines.

ELIGIBILITY:
Inclusion Criteria:

* Patient with pathologically proven diagnosis of adenocarcinoma of the pancreas
* After chemotherapy, tumor is determined to be either locally advanced or unresectable by hepatobiliary surgeon; or tumor is considered potentially resectable but subject does not proceed with surgical resection for any reason
* Have completed first line chemotherapy without progression or non-regional metastases
* Tumor is radiographically evident on CT scan after chemotherapy
* Tumor is anatomically amenable to SBRT, e.g. does not directly invade the stomach or bowel
* Tumor is amenable to intra-tumor injection under endoscopic ultrasound guidance
* ECOG performance status 0-2
* Patients with childbearing potential must demonstrate a negative urine or serum pregnancy test
* Male or female subjects, aged at least 18 years; Female subjects of childbearing potential may participate if adequate contraception is used during, and for at least the three months after study completion; Male subjects with partners of childbearing potential may participate in the study if they had a vasectomy at least 6 months prior to randomization or if adequate contraception is used during, and for at least the three months after study completion; Adequate contraception is defined as resulting in a failure rate of less than 1% per year
* Patient must be able to understand and willingly sign study specific informed consent prior to study entry
* Anticipated life expectancy ≥ 12 weeks
* Patients aged at least 18 years of age

Exclusion Criteria:

* Progression of disease or metastatic disease after first line systemic therapy
* Prior radiation treatment or surgical resection of any pancreatic malignancy
* Inability to tolerate SBRT, Endoscopic ultrasound or IL-12 Injection procedure
* Lack of radiographically evident disease after first line chemotherapy
* Severe, active comorbidity that shortens the patient's life expectancy to less than 12 weeks
* History of past malignancy
* Patient who is pregnant and/or breastfeeding
* Inability to comply with other required protocol procedures including required biopsies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2026-12-01 (Estimated); Primary Completion 2028-12 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability]) | 3 years
  The Primary objective of the safety lead in component is to report acute, attributable, gastrointestinal toxicity
Maximum tolerable dose [Safety and Tolerability] | 3 years
  Maximum tolerable dose is defined by less than or equal to 30% dose limiting toxicity (DLT) event rate within a given dose

SECONDARY OUTCOMES:
Rate of radiographic response | 2 months
  This study will assess radiographic response following SBRT and PCX12 utilizing RECIST 1.1 criteria
Change in biomarkers of innate and adaptive immunity | baseline and 4 weeks
  A combination of flow/mass cytometry will be employed to assess intratumoral immune cells before and after treatment. Specifically, cells of the adaptive immune system, namely B and T cells (both CD4+ and CD8+), along with innate cells including monocytes, macrophages, neutrophils, and natural killer cells will be investigated and percent of total CD45+ cells along with absolute cell number will be tabulated. Additionally, markers of activation (IFNg, TNF, etc.) along with suppression (PD1, PD-L1, LAG3, etc.) will be included in the panel of analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Haoming Qiu, Principal Investigator — University of Rochester
Locations (1):
- University of Rochester, Rochester, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided